CLINICAL TRIAL: NCT06269393
Title: An Exploratory Study of the Efficacy and Safety of IBI311, a Modified Anti-IGF-1R Antibody, in Patients With Steroid-resistant, Thyroid Associated Ophthalmopathy
Brief Title: A Study of IBI311 in Subjects With Steroid-resistant, Thyroid Associated Ophthalmopathy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Xiuying, associate chief physician, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI311Y101
Record Dates: First submitted 2024-01-25; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Thyroid Associated Ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants with TAO will be randomized to receive 4 intravenous infusions of placebo with an interval of 3 weeks, followed by 4 intravenous infusions of IBI311 with an interval of 3 weeks.
  Interventions: Drug: Placebo
- IBI311 (Active Comparator): Participants with TAO will be randomized to receive 8 intravenous infusions of IBI311 with an interval of 3 weeks.
  Interventions: Drug: IBI311

INTERVENTIONS:
Drug: Placebo — Placebo group: 10 mg/kg of placebo on Day 1, followed by 20 mg/kg, q3W of placebo for the following 3 infusions.10 mg/kg of IBI311 at Week 12, followed by 20 mg/kg, q3W of IBI311 for the remaining 3 infusions.
  Arms: Placebo
Drug: IBI311 — IBI311 group: 10 mg/kg of IBI311 on Day 1, followed by 20 mg/kg, q3W of IBI311 for the remaining 7 infusions; .
  Arms: IBI311

SUMMARY:
This is an exploratory study of the efficacy and safety of IBI311, a modified anti-IGF-1R antibody, in patients with steroid-resistant, thyroid associated ophthalmopathy (TAO). This study includes two stages. Stage I is a single-center, single-arm, open-label clinical study designed to evaluate the safety and tolerability of IBI311 in subjects with TAO. Approximately 10 subjects meeting the study eligibility criteria will be enrolled. Stage II is a single-center, randomized, double-masked, placebo-controlled clinical trial designed to evaluate the efficacy and safety of IBI311 in subjects with steroid-resistant TAO. Approximately 54 subjects meeting the study eligibility criteria will be randomly assigned to IBI311 or placebo on day 1 (D1) in a 2:1 ratio stratified by disease activity.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Male or female subject between 18 and 80 years (inclusive) at Screening.
3. Steroid-resistant TAO, defined as poor response to steroid after completing a 3-month steroid pulse therapy (4.5g to 8.0g methylprednisolone) or 3-6 months of oral glucocorticoids treatment (i.e., CAS decreased by < 2 points, or proptosis decreased by < 2mm, or no improvement in diplopia), or relapse of TAO after steroid withdrawal (CAS increased by ≥2 points and CAS≥3 points [7-item scale] in either eye, or proptosis increased by ≥2 mm, or Gorman diplopia score increased by ≥1 point).
4. Moderate-to-severe active TAO or chronic TAO at screening:

   Inclusion criteria for subjects with moderate-to-severe active TAO:
   * Active TAO, with CAS ≥3 in the study eye during the screening period;
   * Proptosis ≥18 mm in the study eye;
   * Moderate to severe active TAO, usually associated with at least two of the following manifestations: eyelid retraction ≥ 2 mm, moderate or severe soft tissue involvement, proptosis ≥ 3 mm above upper limit of normal (ULN), inconstant or constant diplopia (Gorman subjective diplopia score 2-3);

   Inclusion criteria for subjects with chronic TAO:
   * CAS ≤2 in both eyes during the screening period;
   * Proptosis ≥18 mm in the study eye;
   * A clinical diagnosis of chronic non-active TAO at screening was defined as CAS ≤2 in both eyes for at least 6 months prior to screening, or having all of the following characteristics: no progression of proptosis, no newly onset diplopia or diplopia progression induced by TED at least 6 months prior to screening, and no new inflammatory TAO symptoms.
5. Infertile female subjects or fertile female subjects with negative blood pregnancy test results during the screening period and agrees to take contraceptive measures from screening to 120 days after the last dose; male subjects should agree to use contraceptive measures from screening to 120 days after the last dose.

Exclusion Criteria:

Subjects will be ineligible for study participation if they meet any of the following criteria:

1. Decreased best-corrected visual acuity due to optic neuropathy (defined as a ≥ 2-line decrease in best-corrected visual acuity due to optic neuropathy within the past 180 days), newly emerging visual field defects or color vision impairment secondary to optic nerve damage;
2. Subjects with corneal ulcer;
3. Immediate orbital radiotherapy or orbital decompression as judged by investigators;
4. Orbital radiation therapy or surgical treatment for TAO, including orbital decompression, strabismus diorthosis and eyelid diorthosis, at any time before baseline, or planned to have the aforementioned treatments during the study;
5. Subjects with poorly controlled thyroid function, defined as FT3 or FT4 levels deviating from the normal reference ranges of the local study site laboratories by more than 50% at screening;
6. Receiving Teprotumumab or IBI311 at any time before baseline;
7. Receiving anti-CD20 antibody or interleukin-6 receptor antibody treatment within 180 days prior to baseline;
8. Oral or intravenous administration of any other non-steroid immunosuppressant within 90 days prior to baseline

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
The proptosis responder rate (defined as percentage of subjects with a ≥ 2mm reduction from baseline in proptosis in the study eye, without deterioration [≥ 2 mm increase] of proptosis in the non-study eye) of the study eye. | Week 12
  Proptosis assessment: proptosis of the study eye as measured by Hertel exophthalmometer.

SECONDARY OUTCOMES:
Overall responder rate in proptosis of the study eye. | Weeks 12 and 24
  Proptosis assessment: proptosis of the study eye as measured by Hertel exophthalmometer.
Percentage of subjects with a CAS value of 0 or 1 | Weeks 12 and 24
  CAS Assessment Form
Diplopia responder rate (defined as percentage of subjects with a ≥ 1-grade improvement in diplopia) | Weeks 12 and 24
  Gorman subjective diplopia score.

OTHER OUTCOMES:
Safety and tolerability of intravenous IBI311 in subjects with TAO | Up to 24 weeks
  Incidence, severity, relatedness to the study drug, etc. of ocular and systemic adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Wenhui Ren, Principal Investigator — Peking University People's Hospital Research Office
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China